CLINICAL TRIAL: NCT00131300
Title: A Study of the Safety and Efficacy of Synvisc in Patients With Symptomatic Shoulder Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNV-002-01
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis; Musculoskeletal Diseases
Keywords: Osteoarthritis of the shoulder; Musculoskeletal
MeSH Terms: conditions — Osteoarthritis; Musculoskeletal Diseases

INTERVENTIONS:
Device: Synvisc (hylan G-F 20)

SUMMARY:
This clinical study is to evaluate the safety and efficacy of Synvisc in patients with symptomatic shoulder osteoarthritis (OA). Patients will be given Synvisc, with the possible administration of a second injection where insufficient symptomatic pain relief was experienced during the 3 month follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic OA pain of shoulder (gleno-humeral)

Exclusion Criteria:

* Patients with current or prior conditions or treatment that would impede measurement of efficacy or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-04; Study Completion 2006-02

PRIMARY OUTCOMES:
Pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- France (4):
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Clinique Saint Anne Lumiere, Lyon
  - Centre de Medecine et Traumatologie du Sport Clinique du Sport, Mérignac
  - CHRU Hopital Trousseau, Tours
- Germany (2):
  - August-Viktoria-Klinik, Bad Oeynhausen
  - Universitatsklinik und Poliklinik Orthopadie & Physikalische Medizin, Halle